CLINICAL TRIAL: NCT01536288
Title: Can Rhodiola Crenulata Intake Improve Oxygen Saturation and Decrease the Incidence of Acute Mountain Sickness.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: NSC 99-3114-B-182A-002
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2011-11

CONDITIONS: Acute Mountain Sickness; Environmental Illness
Keywords: acute mountain sickness; AMS; Rhodiola Crenulata; mountaineering; pulse oximetry; oxygen saturation
MeSH Terms: conditions — Altitude Sickness; Environmental Illness | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rhodiola crenulata-placebo sequence (Active Comparator): Rhodiola crenulata for the first treatment period and placebo for the second treatment period, with a washout period of 4 months. Overall study population were 120 subjects, who were randomised and allocated into 2 sequences.
  Interventions: Drug: Rhodiola crenulata; Drug: placebo
- Placebo-Rhodiola crenulata sequence (Active Comparator): Placebo for the first treatment period and Rhodiola crenulata for the second treatment period, with a washout period of 4 months. Overall study population were 120 subjects, who were randomised and allocated into 2 sequences.
  Interventions: Drug: Rhodiola crenulata; Drug: placebo

INTERVENTIONS:
Drug: Rhodiola crenulata — Rhodiola crenulata:capsules, 800 mg daily for 7 days before ascent and 2 days during mountaineering
  Other Names: Rhodiola; Golden root; Hong Jing Tian
Drug: placebo — Placebo:capsules, 800 mg daily for 7 days before ascent and 2 days during mountaineering
  Other Names: Starch

SUMMARY:
Traditional folk medicine in the Arctic and Himalayan areas used Rhodiola species to enhance physical endurance, prevent aging, resist acute mountain sickness (AMS), and to treat fatigue, depression, anemia, impotence and respiratory infections. Rhodiola crenulata are widely used to prevent AMS in Himalayan areas and Lhasa in Tibet but none was examined by human study. The investigators conducted a randomized, double blind, placebo controlled, crossover study to investigate the efficacy of Rhodiola crenulata in preventing AMS.

DETAILED DESCRIPTION:
The number of people traveling to altitude for work or for recreation is rising, and increased media attention towards these activities has also raised the profile of altitude related illness. The most effective preventive measure for acute mountain sickness (AMS)-gradual ascent-is frequently difficult or impractical for modern international travel to locations such as Lhasa in Tibet (3650 m) and La Paz in Bolivia (3740 m). In order to solve this problem, prophylactic acetazolamide was most commonly used. But prescription needed and side effects such as paresthesia and nausea are the disadvantage of using acetazolamide. Some over-the-counter herbal supplements with essentially no adverse effect were widely used, such as Rhodiola species. Rhodiola crenulata are widely used to prevent AMS in Himalayan areas and Lhasa in Tibet but none was examined by human study. The investigators conducted a randomized, double blind, placebo controlled, crossover study to investigate the efficacy of Rhodiola crenulata in preventing AMS.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 55 years.
* able to complete the study protocol of 9-day study regimens and mountain climbing twice.
* no prophylactic medication or herb one month before ascent.
* maintaining the same living conditions and habits four months before the first mountain climbing and four months between two mountaineering.

  * living in the same altitude or within a difference of 200 meters.
  * no additional physical training.
  * no plan to gain or loss weight.
  * no altitude exposure above 2500m.

Exclusion Criteria:

* any history of chronic obstructive pulmonary disease, heart failure, cerebral neoplasm, mania, renal or hepatic insufficiency.
* women in pregnancy or intending of pregnancy during the 4-month study period.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Incidence measured by Lake Louise acute mountain sickness score (LLS) ≥ 3 with headache and one other symptom. | within 18 hours after ascent to altitude 3100m
  The LLS rates 5 symptoms (headache, gastrointestinal symptoms such as nausea and vomiting, fatigue and/or weakness, dizziness and/or light-headedness, and difficulty sleeping), with each item graded on a scale from 0 to 3. A score of 3 points or greater constitutes AMS.

SECONDARY OUTCOMES:
blood oxygen content | on arrival of altitude 3100m
  Blood oxygen content was measured by pulse oximetry (NPB 40, Nellcor, Pleasanton, CA, USA) within 1-2 hours after ascent to altitude 3100m.
severe AMS | within 18 hours after ascent to altitude 3100m
  Incidence measured by Lake Louise acute mountain sickness score (LLS) ≥ 5 with headache and one other symptom.
severity of headache, incidence of headache and severe headache | Within 18 hours after ascent to altitude 3100m
  severe headache is determined by cut off between scores of 1 and 2 on the Lake Louise survey (ascending scale of 0-3 for severity)

CONTACTS AND LOCATIONS:
Overall Officials: Te-Fa Chiu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Dept of Emergency medicine, Chang Gung Memorial Hospital, Kweishan, Taoyuan, Taiwan

REFERENCES:
- [Background] Hackett PH, Roach RC. High-altitude illness. N Engl J Med. 2001 Jul 12;345(2):107-14. doi: 10.1056/NEJM200107123450206. No abstract available. PMID 11450659
- [Background] Imray C, Booth A, Wright A, Bradwell A. Acute altitude illnesses. BMJ. 2011 Aug 15;343:d4943. doi: 10.1136/bmj.d4943. No abstract available. PMID 21844157
- [Background] Chow T, Browne V, Heileson HL, Wallace D, Anholm J, Green SM. Ginkgo biloba and acetazolamide prophylaxis for acute mountain sickness: a randomized, placebo-controlled trial. Arch Intern Med. 2005 Feb 14;165(3):296-301. doi: 10.1001/archinte.165.3.296. PMID 15710792
- [Background] Hackett PH, Rennie D, Levine HD. The incidence, importance, and prophylaxis of acute mountain sickness. Lancet. 1976 Nov 27;2(7996):1149-55. doi: 10.1016/s0140-6736(76)91677-9. PMID 62991
- [Background] Zell SC, Goodman PH. Acetazolamide and dexamethasone in the prevention of acute mountain sickness. West J Med. 1988 May;148(5):541-5. PMID 3051673
- [Background] Dumont L, Mardirosoff C, Tramer MR. Efficacy and harm of pharmacological prevention of acute mountain sickness: quantitative systematic review. BMJ. 2000 Jul 29;321(7256):267-72. doi: 10.1136/bmj.321.7256.267. PMID 10915127
- [Background] Basnyat B, Gertsch JH, Holck PS, Johnson EW, Luks AM, Donham BP, Fleischman RJ, Gowder DW, Hawksworth JS, Jensen BT, Kleiman RJ, Loveridge AH, Lundeen EB, Newman SL, Noboa JA, Miegs DP, O'Beirne KA, Philpot KB, Schultz MN, Valente MC, Wiebers MR, Swenson ER. Acetazolamide 125 mg BD is not significantly different from 375 mg BD in the prevention of acute mountain sickness: the prophylactic acetazolamide dosage comparison for efficacy (PACE) trial. High Alt Med Biol. 2006 Spring;7(1):17-27. doi: 10.1089/ham.2006.7.17. PMID 16544963
- [Background] Imray C, Wright A, Subudhi A, Roach R. Acute mountain sickness: pathophysiology, prevention, and treatment. Prog Cardiovasc Dis. 2010 May-Jun;52(6):467-84. doi: 10.1016/j.pcad.2010.02.003. PMID 20417340
- [Background] Leadbetter G, Keyes LE, Maakestad KM, Olson S, Tissot van Patot MC, Hackett PH. Ginkgo biloba does--and does not--prevent acute mountain sickness. Wilderness Environ Med. 2009 Spring;20(1):66-71. doi: 10.1580/08-WEME-BR-247.1. PMID 19364166
- [Background] Gertsch JH, Basnyat B, Johnson EW, Onopa J, Holck PS. Randomised, double blind, placebo controlled comparison of ginkgo biloba and acetazolamide for prevention of acute mountain sickness among Himalayan trekkers: the prevention of high altitude illness trial (PHAIT). BMJ. 2004 Apr 3;328(7443):797. doi: 10.1136/bmj.38043.501690.7C. Epub 2004 Mar 11. PMID 15070635
- [Background] Gertsch JH, Seto TB, Mor J, Onopa J. Ginkgo biloba for the prevention of severe acute mountain sickness (AMS) starting one day before rapid ascent. High Alt Med Biol. 2002 Spring;3(1):29-37. doi: 10.1089/152702902753639522. PMID 12006162
- [Background] van Patot MC, Keyes LE, Leadbetter G 3rd, Hackett PH. Ginkgo biloba for prevention of acute mountain sickness: does it work? High Alt Med Biol. 2009 Spring;10(1):33-43. doi: 10.1089/ham.2008.1085. PMID 19278351
- [Background] Zhang ZJ, Tong Y, Zou J, Chen PJ, Yu DH. Dietary supplement with a combination of Rhodiola crenulata and Ginkgo biloba enhances the endurance performance in healthy volunteers. Chin J Integr Med. 2009 Jun;15(3):177-83. doi: 10.1007/s11655-009-0177-x. Epub 2009 Jul 2. PMID 19568709
- [Background] Tu Y, Roberts L, Shetty K, Schneider SS. Rhodiola crenulata induces death and inhibits growth of breast cancer cell lines. J Med Food. 2008 Sep;11(3):413-23. doi: 10.1089/jmf.2007.0736. PMID 18800886
- [Background] Nakamura S, Li X, Matsuda H, Yoshikawa M. Bioactive constituents from Chinese natural medicines. XXVIII. Chemical structures of acyclic alcohol glycosides from the roots of Rhodiola crenulata. Chem Pharm Bull (Tokyo). 2008 Apr;56(4):536-40. doi: 10.1248/cpb.56.536. PMID 18379104
- [Background] Zheng KY, Guo AJ, Bi CW, Zhu KY, Chan GK, Fu Q, Xu SL, Zhan JY, Lau DT, Dong TT, Choi RC, Tsim KW. The extract of Rhodiolae Crenulatae Radix et Rhizoma induces the accumulation of HIF-1alpha via blocking the degradation pathway in cultured kidney fibroblasts. Planta Med. 2011 Jun;77(9):894-9. doi: 10.1055/s-0030-1250627. Epub 2010 Dec 14. PMID 21157678
- [Background] Zhao Y, Qi LW, Wang WM, Saxena PK, Liu CZ. Melatonin improves the survival of cryopreserved callus of Rhodiola crenulata. J Pineal Res. 2011 Jan;50(1):83-8. doi: 10.1111/j.1600-079X.2010.00817.x. Epub 2010 Nov 15. PMID 21073518
- [Background] Lee OH, Kwon YI, Apostolidis E, Shetty K, Kim YC. Rhodiola-induced inhibition of adipogenesis involves antioxidant enzyme response associated with pentose phosphate pathway. Phytother Res. 2011 Jan;25(1):106-15. doi: 10.1002/ptr.3236. PMID 20623718
- [Background] Li T, Zhang H. Identification and comparative determination of rhodionin in traditional tibetan medicinal plants of fourteen Rhodiola species by high-performance liquid chromatography-photodiode array detection and electrospray ionization-mass spectrometry. Chem Pharm Bull (Tokyo). 2008 Jun;56(6):807-14. doi: 10.1248/cpb.56.807. PMID 18520085
- [Background] Li T, Zhang H. Application of microscopy in authentication of traditional Tibetan medicinal plants of five Rhodiola (Crassulaceae) alpine species by comparative anatomy and micromorphology. Microsc Res Tech. 2008 Jun;71(6):448-58. doi: 10.1002/jemt.20570. PMID 18300292
- [Background] Kwon YI, Jang HD, Shetty K. Evaluation of Rhodiola crenulata and Rhodiola rosea for management of type II diabetes and hypertension. Asia Pac J Clin Nutr. 2006;15(3):425-32. PMID 16837437
- [Background] Panossian A, Wikman G, Sarris J. Rosenroot (Rhodiola rosea): traditional use, chemical composition, pharmacology and clinical efficacy. Phytomedicine. 2010 Jun;17(7):481-93. doi: 10.1016/j.phymed.2010.02.002. Epub 2010 Apr 7. PMID 20378318
- [Background] Wang S, Wang FP. [Studies on the chemical components of Rhodiola crenulata]. Yao Xue Xue Bao. 1992;27(2):117-20. Chinese. PMID 1414365
- [Background] Wang S, You XT, Wang FP. [HPLC determination of salidroside in the roots of Rhodiola genus plants]. Yao Xue Xue Bao. 1992;27(11):849-52. Chinese. PMID 1300030
- [Background] Wang SH, Chen YC, Kao WF, Lin YJ, Chen JC, Chiu TF, Hsu TY, Chen HC, Liu SW. Epidemiology of acute mountain sickness on Jade Mountain, Taiwan: an annual prospective observational study. High Alt Med Biol. 2010 Spring;11(1):43-9. doi: 10.1089/ham.2009.1063. PMID 20367488
- [Background] Karinen HM, Peltonen JE, Kahonen M, Tikkanen HO. Prediction of acute mountain sickness by monitoring arterial oxygen saturation during ascent. High Alt Med Biol. 2010 Winter;11(4):325-32. doi: 10.1089/ham.2009.1060. PMID 21190501
- [Background] Roach RC, Greene ER, Schoene RB, Hackett PH. Arterial oxygen saturation for prediction of acute mountain sickness. Aviat Space Environ Med. 1998 Dec;69(12):1182-5. PMID 9856544
- [Background] Jackson SJ, Varley J, Sellers C, Josephs K, Codrington L, Duke G, Njelekela MA, Drummond G, Sutherland AI, Thompson AA, Baillie JK. Incidence and predictors of acute mountain sickness among trekkers on Mount Kilimanjaro. High Alt Med Biol. 2010 Fall;11(3):217-22. doi: 10.1089/ham.2010.1003. PMID 20919888
- [Derived] Chiu TF, Chen LL, Su DH, Lo HY, Chen CH, Wang SH, Chen WL. Rhodiola crenulata extract for prevention of acute mountain sickness: a randomized, double-blind, placebo-controlled, crossover trial. BMC Complement Altern Med. 2013 Oct 31;13:298. doi: 10.1186/1472-6882-13-298. PMID 24176010
- See also: International society of mountain medicine — http://www.ismmed.org/
- See also: Acute mountain sickness, Kingnet, national web hospital — http://hospital.kingnet.com.tw/essay/essay.html?category=%C2%E5%C3%C4%AFe%AFf&pid=13719
- See also: American college emergency physicians — http://www.acep.org/
- See also: wilderness medicine, medicine and the spirit of adventure — http://www.wilderness-medicine.com/